CLINICAL TRIAL: NCT07145645
Title: Topical Diclofenac vs. Oral Ibuprofen for Musculoskeletal Pain in Children: A Multi-centre, Randomized Pilot Feasibility Trial
Brief Title: Topical Diclofenac vs.Oral Ibuprofen for MSK Pain in Children
Acronym: TOP-MAP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOPMAP-25-02-2025
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: Musculoskeletal Injury; Pediatrics; Sprain and Strain of Ankle; Sprain Knee; Strain Knee
Keywords: Non Steroidal Anti-Inflammatory; Pediatric Emergency Department; Pediatrics; Ankle or Knee Injury; Topical NSAIDs
MeSH Terms: conditions — Sprains and Strains; Knee Injuries | interventions — diclofenac diethylamine

STUDY DESIGN:
Intervention Model Description: This is a pilot study to determine the feasibility of a large, multi-centre, non-inferiority trial of topical vs oral NSAIDs for acute pediatric MSK injuries. Both study medications (topical and oral) will be administered simultaneously to maintain masking of participants and accuracy of pain assessments. Medication will be given three times daily for the first 72 hours, followed by as-needed dosing for a total of 14 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The double-dummy design is used since the two medications (oral vs. topical) look very different. Participants will take both medications at each time point (one being active and one being placebo) to maintain masking of the participants. The oral medication and the topical medication are provided to the participants in identical packaging to maintain blinding. Only the pharmacists will know which group the participant is in. If there's a medical reason to find out (for example, if the participant has a rare or unexpected allergic reaction), the doctors can access that information immediately.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active topical Diclofenac Diethylamine emulgel (Experimental): Topical Diclofenac emulgel is a topical NSAID with clinically proven analgesic, anti-inflammatory and antipyretic properties when applied directly to a soft tissue injury. NSAIDs reduce pain principally by inhibiting formation of prostaglandins, leukotrienes and free oxygen radicals. Diclofenac can be expected to produce a direct anti-inflammatory and analgesic effect to the area applied.
  Participants randomized to the experimental arm will be given topical diclofenac gel (11.6 mg/g). Dosing is based on the following weight bands:
  25 kg: 2 grams/dose;
  ≥25 kg - <40 kg: 3 grams/dose; and >40 kg: 4 grams/dose.
  Interventions: Drug: Voltaren Topical Gel; Drug: ORA-Blend Oral Suspension
- Active Ibuprofen suspension (Active Comparator): Active oral ibuprofen suspension. The ibuprofen suspension dose is 10 mg/kg to a maximum of 600 mg. Ibuprofen is commonly used in ED's as usual care for treatment of soft tissue injuries in pediatric patients.
  Interventions: Drug: Ibuprofen Oral Suspension 100 mg/5mL; Drug: VersaPro Cream Base for Compounding

INTERVENTIONS:
Drug: Voltaren Topical Gel — Topical diclofenac emulgel (Voltaren) 11.6 mg/g. Dosing is based on weight bands: 25 kg: 2 grams/dose, ≥25 kg - <40 kg: 3 grams/dose; and >40 kg: 4 grams/dose. ATC code: M02A A15.
  Other Names: diclofenac emulgel; diclofenac diethylamine
  Arms: Active topical Diclofenac Diethylamine emulgel
Drug: Ibuprofen Oral Suspension 100 mg/5mL — Children's Ibuprofen Oral suspension (Motrin) 100mg/5 mL . Dosing is 10 mg/kg to a maximum of 600mg.
  Other Names: Children's Motrin; Ibuprofen Oral Suspension
  Arms: Active Ibuprofen suspension
Drug: ORA-Blend Oral Suspension — Oral Ibuprofen suspension (labelled as ibuprofen) given at 10 mg/kg to a maximum of 600mg each dose.
  Arms: Active topical Diclofenac Diethylamine emulgel
Drug: VersaPro Cream Base for Compounding — Topical Versapro Cream emulgel (labeled as diclofenac diethylamine). Dose is based on the following weight bands: 25 kg: 2 grams/dose;
  ≥25 kg - <40 kg: 3 grams/dose; and >40 kg: 4 grams/dose.
  Other Names: Versapro Gel
  Arms: Active Ibuprofen suspension

SUMMARY:
The TOP-MAP pilot trial has multiple goals. The first goal of this pilot clinical trial is to find out if it will be possible to carry out a study at multiple pediatric emergency department sites (Peds ED) comparing Non-Steroidal Anti-Inflammatory (NSAID) gel applied to a new ankle or knee injury to NSAIDs taken by mouth in kids aged 6-18. The investigators want to determine if the gel works as well or better at reducing pain than NSAIDs given by mouth. Based on studies done on adults, the investigators know that NSAIDs that are applied directly to an injury work as well at relieving pain as NSAIDs that are taken by mouth. Another goal of this pilot trial is to determine if it is possible to recruit participants to the study, and if the participants complete the questionnaire and take the medications as prescribed on Day 1.

The participants will be in the study for 14 days. Participants will be required to take the oral NSAID medication and to apply the topical NSAID gel 3 times a day for the first 3 days after their visit to the ED. The investigators will ask the participants to rate their pain on a scale of 0 (no pain) to 10 (worst pain ever) before and after they use the medicine. On day 7, the participants will rate their pain, and their activity level. On day 14 participants will do the same.

DETAILED DESCRIPTION:
In Canada, musculoskeletal sprains and strains account for 10% of Emergency department visits in children aged 10-17 years of age. Unlike upper limb injuries, which are often fractured, injuries to the ankle and knees are non-fractured soft tissue injuries in 88% and 91% respectively. Management of such injuries is focused on pain and inflammation management through pharmacotherapy, cryotherapy and early mobilization while avoiding casting.

Oral ibuprofen, a non-steroidal anti-inflammatory drug (NSAID) is the recommended first-line pharmacotherapy for mild to moderate musculoskeletal (MSK) injury related pain. However, alternatives such as topical NSAIDs (e.g., diclofenac emulgel) are commonly recommended in adults. Among adults their effect is equivalent to oral NSAIDs and they can be directly applied to the injured area resulting in a lower risk of systemic adverse events (AE's). Despite their frequent use in adults, topical NSAIDs are currently not recommended for children due to a lack of supporting data.

Based on adult data, the investigators hypothesize that topical NSAIDs provide similarly effective pain management to oral NSAIDs in children with acute MSK injuries with a reduced risk of systemic AEs. This pilot trial will assess the feasibility of a definitive non-inferiority trial of topical diclofenac emulgel vs. oral ibuprofen for children with acute ankle or knee soft tissue injuries. The results of a definitive trial have the potential to alter current pediatric MSK injury management if topical diclofenac emulgel is indeed non-inferior to oral ibuprofen for pain relief, with an expected lower risk of systemic AEs.

In children aged 6 to <18 years with an acute (≤4-days) ankle or knee non-fractured soft tissue injury (e.g., sprain, strain or contusion), is topical diclofenac emulgel 11.6 mg/g non-inferior to oral ibuprofen (both administered three times daily) in reducing pain during the 72 hours following ED discharge? This pilot randomized, double-dummy, blinded (participants, clinicians, outcome assessors, investigators), two-centre ED trial will enroll 60 participants, following the 2010 CONSORT statement.

Study medications will be administered simultaneously to maintain masking of participants and accuracy of pain assessments, three times daily for the first 72 hours, followed by as-needed dosing for a total of 14 days.

This pilot will inform the planning of a definitive trial by assessing a) feasibility of recruiting patients in EDs; b) acceptability of interventions; c) ability to collect at-home pain assessments; d) identifying pain assessment time-point with the highest completion and effect; and e) refining sample size calculations from variance around clinical outcomes data. The investigators will evaluate the impact of the eligibility criteria and identify which groups of children are being excluded and why. This data will be used to inform discussions to finalize the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 to 18 years old.
2. Injury less than or equal to 4 days old
3. Non-fractured MSK soft-tissue injury (ankle or knee, confirmed clinically and/or radiographically)
4. Pain score of more than or equal to 3 on the verbal numerical rating scale, with movement in the past 2 hours or before analgesia

Exclusion Criteria:

1. Previous enrolment in the trial
2. Barriers to topical treatment application, including skin conditions (e.g. eczema, infection, open wounds) or overlying material (e.g., rigid cast) which would make applying topical treatment impossible.
3. Any other history, condition, therapy, or uncontrolled intercurrent illness, which could, in the opinion of the Qualified Medical Investigator or treating physician, would make the participant unsuitable for this study
4. Any contraindication to NSAID use including but not limited to a history of GI bleeding, gastric ulcer, inflammatory bowel disease, prior cerebrovascular bleeding, bleeding diathesis, interstitial kidney disease
5. Taking NSAIDs daily for other indications (e.g, chronic pain or arthritis)
6. Known hypersensitivity to ibuprofen, diclofenac or other NSAIDs.
7. Any known allergy or intolerance to any components (e.g., aloe vera) included in the oral or topical preparations of the investigational products
8. Current use of prohibited medications known to impair renal function when combined with NSAIDs or cause potential additive risks of gastrointestinal toxicity and renal impairment
9. Absence of a parent/guardian for children who are not mature minors.
10. Caregiver and/or child cognitive impairment precluding the ability to complete study procedures
11. Inability to obtain consent, and to complete follow-up surveys due to language barrier
12. Known or suspected late pregnancy (gestational age ≥20 weeks) at the time of enrolment or breastfeeding females, due to the risk of premature closure of the ductus arteriosus associated with NSAID use
13. Current enrollment in another pain-related clinical trial or in a study that, in the opinion of the Qualified Medical Investigator, may interfere with enrollment, involve investigational products that interact with study medications, or compromise follow-up and outcome assessment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a large trial to be measured by the following: 1. 50% consent rate from all eligible candidates approached; 2. Achieve 80% completion rate of the first 24 hour survey, 3. Achieve 80% adherence rate to Day 1 dosing regimen. | Will be evaluated at study end, 18 months.
  To determine the feasibility of conducting a large multi-centre non-inferiority trial. This will be evaluated with the use of descriptive statistics of the following three measurements:
  1. The investigators aim to achieve a 50% consent rate from all eligible candidates approached to participate.
  2. The investigators' goal is to have 80% of the consented and enrolled participants complete the Day 1 (first 24-hour survey) follow up survey. This will be measured by counting the number of completed Day 1 surveys out of all Day 1 surveys that are expected to be completed.
  3. The third metric is to have 80% of the participants adhere to the dosing regimen in the first 24 hours after discharge from the ED. This will be measured by calculating the number of participants that administered all 3 doses of study medications in the first 24 hours.

SECONDARY OUTCOMES:
Pain relief as measured on the verbal Numerical Rating scale. | First 24 hours after ED discharge
  To assess between group mean differences in reported pain scores as measured on the 11-point verbal numerical scale. The vNRS is scaled from 0 (no pain) to 10 (worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Eltorki, MBChB, MSc, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: Yes
De-identified, anonymized data that give support to the results reported in the study may be shared with other researchers. Any data that could potentially identify participants due to a low N (ie; race data reported of less than 5) will not be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Requests to access data can be made 9 months after the publication, for 36 months following article publication.
Access Criteria: Proposals to access the anonymized, deidentified data should be submitted to the Principal Investigator, Dr. Mohamed Eltorki (mmeltork@ucalgary.ca). Only those researchers who submit a methodologically sound proposal to use the data for a meta-analysis will be considered for access.

REFERENCES:
- [Background] ChildHealth BC. Children's Emergency Department Services. Vancouver, BC: Child Health BC,2020/07/20. (Acessed 2024-08-07, athttps://www.childhealthbc.ca/sites/default/files/20-07-01-ed-tiers-setting-the-stage-1819-data.pdf.)
- [Background] Wang C, Toigo S, Zutrauen S, McFaull SR, Thompson W. Injuries among Canadian children and youth: an analysis using the 2019 Canadian Health Survey on Children and Youth. Health Promot Chronic Dis Prev Can. 2023 Feb;43(2):98-102. doi: 10.24095/hpcdp.43.2.05. PMID 36794826